CLINICAL TRIAL: NCT03929276
Title: Efficacy of High-intensity Laser Therapy in Patients With Adhesive Capsulitis
Brief Title: Laser Therapy in Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Tuğba Atan, Assoc. Prof., Hitit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-KAEK-061
Record Dates: First submitted 2019-04-22; First posted 2019-04-26 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: adhesive capsulitis; high-intensity laser therapy
MeSH Terms: conditions — Bursitis | interventions — Exercise Therapy; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high-intensity laser therapy & exercises (Experimental): High-intensity laser therapy application with iLux Laser device + exercise program
  Interventions: Device: high-intensity laser therapy & exercises; Other: exercise
- Shame laser & exercises (Placebo Comparator): Sham high-intensity laser therapy application with iLux Laser device + exercise program
  Interventions: Device: Shame laser & exercises; Other: exercise
- control - exercises only group (Active Comparator): exercise program
  Interventions: Other: exercise

INTERVENTIONS:
Device: high-intensity laser therapy & exercises — A total of 15 sessions of high-dose laser treatment- i Lux Laser (Mectronic Medicale, Italy)- (in the first phase, 8 Watt for the analgesic effect; in the second phase, 12 Watt in burst mode for the biostimulation effect; and finally in the third phase with 8 Watt) will be applied.
  Arms: high-intensity laser therapy & exercises
Device: Shame laser & exercises — Sham laser treatment (the same device to be used, 0 watts) will be given.
  Arms: Shame laser & exercises
Other: exercise — Therapeutic exercises All participants received 25-minutes of passive stretching, active assisted range of motion and codman pendicular exercises (10 repetitions, 3 sets, 3-minutes rest between sets) to the shoulder joint, supervised by the same physiotherapist five times a week for 3 weeks.

SUMMARY:
Adhesive capsulitis is an idiopathic disease characterized by a decrease in the volume of the glenoid capsule, the development of fibrosis and a progressive decrease in the range of joint movement with pain. Shoulder pain and stiffness are accompanied by disability. The purpose of the study is to evaluate and compare the effects of high-intensity laser therapy on pain, disease - related disability and quality of life in patients with shoulder restriction and pain due to adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis is an idiopathic disease characterized by a decrease in the volume of the glenoid capsule, the development of fibrosis and a progressive decrease in the range of joint movement with pain. Shoulder pain and stiffness are accompanied by disability. It is thought that the incidence is 3% to 5% in the general population and 20% in people with diabetes. Although usually reported to be self-limiting in 2 to 3 years, studies have reported that 40% of patients have persistent pain and stiffness for more than 3 years.

Therefore, various therapies are used to reduce pain and increase the range of motion more rapidly without waiting for spontaneous recovery. Adhesive capsulitis treatment includes conservative and surgical treatment options. The options for non-surgical treatments are pharmacological treatments including intra-articular injection and physical therapy modalities. As for physical therapy modalities, various interventions are used. These include heat or ice, therapeutic ultrasound, transcutaneous electrical nerve stimulation and laser therapies.

The aim of exercise programs consisting of joint range of motion (ROM), strengthening and stretching exercises, proprioceptive neuromuscular facilitation and mobilization techniques is to alleviate pain caused by the capsular contracture and to improve glenohumeral ROM.

The purpose of the study is to evaluate and compare the effects of high-intensity laser therapy on pain, disease - related disability and quality of life in patients with shoulder restriction and pain due to adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with adhesive capsulitis diagnosis by physical examination (Compared with intact side, there is more than 25% limitation in at least two directions of shoulder range of motion)
* Subjects have complaints for at least 1 month
* No pregnancy / breastfeeding

Exclusion Criteria:

* History of bilateral adhesive capsulitis
* History of shoulder trauma, fracture, shoulder shoulder surgery, calcific tendinopathy, glenohumeral osteoarthritis, inflammatory rheumatic diseases, tumor, infection
* History of corticosteroid injection in the shoulder during the last 3 months
* History of recent lung, breast or bypass surgery
* History of cervical radiculopathy / brachial plexus lesion
* History of neuromuscular disease
* History of physical therapy program for the same shoulder in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-09-22 (Actual); Study Completion 2019-09-22 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale for pain (VAS- pain) | 2 weeks
  Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity.

SECONDARY OUTCOMES:
Shoulder pain and disability index | 2 weeks
  It is a self-administered questionnaire and two dimensions are measured, one for pain and the other for functional activities. Scores range from 0 to 100 with scores closer to 0 indicating lower (or no) disability and scores closer to 100 indicating greater disability.
Short Form Health Survey 36 (SF-36) | 2 weeks
  Short- form health survey 36 contains 36 items which are used to evaluate the quality of life of patients with chronic pain. It measures eight different domains that address physical functioning, physical role limitation, pain, general health, vitality, social functioning, emotional role limitation and mental health. The score of each domain ranges from 0 (worse quality of life) to 100 (best quality of life).
Range of motion of shoulder joint measurements | 2 weeks
  shoulder flexion, abduction, external rotation and internal rotation

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Atan, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manske RC, Prohaska D. Diagnosis and management of adhesive capsulitis. Curr Rev Musculoskelet Med. 2008 Dec;1(3-4):180-9. doi: 10.1007/s12178-008-9031-6. PMID 19468904
- [Background] Dudkiewicz I, Oran A, Salai M, Palti R, Pritsch M. Idiopathic adhesive capsulitis: long-term results of conservative treatment. Isr Med Assoc J. 2004 Sep;6(9):524-6. PMID 15373308
- [Derived] Atan T, Bahar-Ozdemir Y. Efficacy of high-intensity laser therapy in patients with adhesive capsulitis: a sham-controlled randomized controlled trial. Lasers Med Sci. 2021 Feb;36(1):207-217. doi: 10.1007/s10103-020-03121-z. Epub 2020 Aug 18. PMID 32808147